CLINICAL TRIAL: NCT00781807
Title: Multi-module Rehabilitation for Patients on LVAD Support - Impact on Long-term Outcomes
Brief Title: Rehabilitation and Outcome for Patients on LVAD Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: Deutsche Stiftung für Herzforschung (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Dr. rer.biol. hum. Christiane Kugler, Hannover Medical School, Clinic für Cardiac, Thoracic, Transplantation and Vascular Surgery, Carl-Neuberg-Str. 1, 30625 Hannover, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DSfH-Project-No. F/05/08
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Exercise Capacity; Quality of Life
Keywords: Heart-Assist-Devices; Rehabilitation; Outcome Assessment (Health Care); Exercise Capacity; Ergometry; Social Support; Quality of Life; Nutrition Assessment; Nutrition Therapy; Neuropsychological Tests
MeSH Terms: interventions — Quality of Life; Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): The prospective intervention group with nutrition management, home-based bicycle ergometer training program and psychosocial support
  Interventions: Other: multi-module rehabilitation program

INTERVENTIONS:
Other: multi-module rehabilitation program — The multi-module rehabilitation program includes:
  1. Nutrition management
  2. Home-based ergometer training program
  3. Psychosocial support
  Other Names: LVAD; long-term support; HRQoL; ergometer training; nutrition management

SUMMARY:
A prospective, multi-module intervention based on nutrition management, psychosocial support, and a controlled home-based physical exercise training program for patients on LVAD- support will be provided to improve outcomes in terms of survival and patients health-related quality of life (HRQoL) for the long-term. Physical capacity, neurocognitive, psychological factors, and adverse events will be assessed as potential independent indicators for HRQoL.

DETAILED DESCRIPTION:
The multi-module intervention program for patients on LVAD support includes nutrition management, home-based ergometer training program, psychosocial support and neurocognitive screening. The nutrition management and physical reconditioning program will be supplemented by psychosocial support targeting the risk of increased stress, anxiety, and depression level. Moreover, standardized neurocognitive screening procedures will be administered to detect neurocognitive dysfunction (except stroke) and will be assessed for their potential to predict limitations in QoL. Adverse events like re-hospitalizations, thromboembolic and bleeding events will be monitored and assessed for their potential to negatively impact QoL.

ELIGIBILITY:
Inclusion Criteria:

* All eligible patients after LVAD implantation for long-term support with follow-up at our outpatient clinic
* Written informed consent
* Sufficient German language skills to read and answer a battery of questionnaires
* 18 years and older

Exclusion Criteria:

* Severe ventricular arrhythmia
* Severe orthopaedic comorbidities
* Illiteracy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-11; Primary Completion 2013-10 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Increase in Quality of Life between hospital discharge after LVAD implant and explantation at least three month | between hospital discharge after LVAD implant and explantation at least three month

SECONDARY OUTCOMES:
Anxiety and depression scores | between hospital discharge after LVAD implant and explantation at least three month
Maximum exercise capacity | between hospital discharge after LVAD implant and explantation at least three month
Body mass index | between hospital discharge after LVAD implant and explantation at least three month
Neurologic events | between hospital discharge after LVAD implant and explantation at least three month
Adverse events | between hospital discharge after LVAD implant and explantation at least three month

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Kugler, Principal Investigator — Hannover Medical School
Locations (2):
- Germany (2):
  - Hannover Medical School, Clinic for Cardiac, Thoracic, Transplantation and Vascular Surgery, Hanover
  - Hannover Medical School, Hanover